CLINICAL TRIAL: NCT05741918
Title: Cardiac Output Measurement in Pediatric Intensive Care Unit by Metabolic Monitor (Fick Method) : Prospective Feasibility Study
Brief Title: Cardiac Output Measurement in Pediatric Intensive Care Unit by Metabolic Monitor (Fick Method) (PEDIA-FICK-ICU)
Acronym: PEDIA-FICK-ICU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RECHMPL22_0227
Record Dates: First submitted 2023-02-13; First posted 2023-02-23 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Intensive Care Units, Pediatric
Keywords: Cardiac output; Oxygen Consumption (VO2); Fick; Pediatric Intensive Care Unit
MeSH Terms: interventions — Echocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pediatric Intensive Care Units Patients (Experimental): Patients under 18 admitted in pediatric intensive care unit
  Interventions: Diagnostic Test: Fick's method; Diagnostic Test: Echocardiography

INTERVENTIONS:
Diagnostic Test: Fick's method — Cardiac output measurement by Fick method
Diagnostic Test: Echocardiography — Cardiac output measurement by echocardiography

SUMMARY:
Cardiac output measurement is one of the most frequently used haemodynamic parameter used for intensive care unit (ICU) patients. In pediatric ICU, it is often measured with echocardiography that is a non-invasive method but is operator dependant and can't provide continuous monitoring.

The goal of this clinical trial is to evaluate the feasibility of cardiac output measurement by Fick's method, non-invasive and allowing continuous monitoring, in comparison to echocardiography in pediatric intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Patient under 18 years old
* Patient over 10 kg
* Patient requiring intubation or intubated with a cuffed tube
* Patient requiring a central venous line in superior vena cava territory

Exclusion Criteria:

* Mechanical ventilation with leak
* Bad echogenicity preventing echocardiography
* Absence of written informed consent
* Patient not affiliated to French Health Insurance or not covered by public health insurance
* Patient with a legal protection

Ages: 28 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2023-08-20 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Intra-class correlation (or concordance) between the measurement of cardiac output (in ml/min) by Fick's method and by echocardiography | Up to day 3

SECONDARY OUTCOMES:
Variations of cardiac output before and after Leg Raise Test | Up to day 3
Adverse events on the day of catheterization | Up to 21 days
  Complications possibly due to Fick's method on the day of catheterization : pneumothorax, bleeding, rhythm disorder, gas embolism, failure to place, other
Adverse events on the day of catheter removal | Up to 21 days
  Complications possibly due to Fick's method on the day of catheter removal : catheter thrombosis, catheter infection, non-functional oximetry catheter

CONTACTS AND LOCATIONS:
Locations (1):
- UH Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No